CLINICAL TRIAL: NCT03581253
Title: Validation of a French-language Version of Specific Quality of Life Questionnaires in Patients With Peripheral Facial Palsy
Brief Title: Validation of a French-language Version of Quality of Life Questionnaires in Patients With Peripheral Facial Palsy
Acronym: PFQDV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-44
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Peripheral Facial Paralysis; Quality of Life
MeSH Terms: conditions — Facial Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- peripheral facial palsy patients (Experimental): peripheral facial palsy patients will performed questionnaires of quality of life ("Facial disability Index" (FDi) and "Facial Clinimetric Evaluation" (FaCE)
  Interventions: Other: Facial disability Index" (FDi); Other: "Facial Clinimetric Evaluation" (FaCE)

INTERVENTIONS:
Other: Facial disability Index" (FDi) — questionnaires regarding to quality of life
Other: "Facial Clinimetric Evaluation" (FaCE) — questionnaires regarding to quality of life

SUMMARY:
Facial palsy is a serious and disabling disease whose drudgery and sensation are probably underestimated. Psychological, social and economic issues have major impacts although vital prognosis is not engaged in this pathology. Facial palsy remains a personal drama for patient. Consequences may take the form of: aesthetic deformation, modification of body image, with socio-professional consequences. Beside unsightly facial aspects, weakness of facial muscles can cause troubles in eating, drinking, talking, communicating personal emotions and communication. Facial palsy impacts patients' quality of life (QOL) and affects mental health. This wide multidimensional concept usually includes self-measures of physical and mental health. QOL is evaluated with general and specific scales. General scales allow to compare QOL of different diseases, when specific scales focus on one disease and consider all aspects related to this disease and therefore are more appropriate and sensitive in dimensions related to patient disease and health.

"Facial disability Index" (FDi) and "Facial Clinimetric Evaluation" (FaCE) are the most used validated questionnaires to assess QOL of patients suffering from peripheral facial palsy (PFP). There is no existing validated questionnaire or scale in French version despite many French studies on PFP available. Using these questionnaires in French language requires translation and strict approval of the new language version. The aim of the study is to translate and validate French versions of specific scales of QOL in peripheral facial palsy patients: FDI and FaCE. Secondary objective is to evaluate QOL of patients depending on PFP etiology. Translation process will be done respecting internationally recognized rules. A pilot study will be performed on 5 physicians and 5 patients in order to validate the questionnaires translations. French versions obtained will be used for their validation on 80 patients suffering from PFP.

Cronbach's alpha will be estimated to check internal consistency of FDI and FaCE scales. Test re-test reliability will be calculated with inter-class correlation, reiterating questionnaires one week later. Scores of FDI and FaCE scales will be compared to other clinical evaluation scales, estimating correlation coefficient. Social function of FDI and FaCE scales will be compared with general scale SF-36 scores, estimating a correlation coefficient.

DETAILED DESCRIPTION:
Facial palsy is a serious and disabling disease whose drudgery and sensation are probably underestimated. Psychological, social and economic issues have major impacts although vital prognosis is not engaged in this pathology. Facial palsy remains a personal drama for patient. Consequences may take the form of: aesthetic deformation, modification of body image, with socio-professional consequences. Beside unsightly facial aspects, weakness of facial muscles can cause troubles in eating, drinking, talking, and communicating personal emotions. Physical as well as psychological repercussions limit daily verbal and non-verbal communication.

Facial palsy impacts patients' quality of life (QOL) and affects mental health. Consequently, QOL impacts and directs the patient's care and the healthcare professionals widely take account of QOL.

This wide multidimensional concept usually includes self-measures of physical and mental health. QOL is evaluated with general and specific scales. General scales allow to compare QOL of different diseases, when specific scales focus on one disease and consider all aspects related to this disease and therefore are more appropriate and sensitive in dimensions related to patient disease and health.

"Facial disability Index" (FDi) and "Facial Clinimetric Evaluation" (FaCE) are the two most used validated questionnaires to assess QOL of patients suffering from peripheral facial palsy (PFP).

There is no existing validated questionnaire or scale in French version evaluating QOL of patients with PFP despite many French studies on PFP available. Using these questionnaires in French language requires translation and strict approval of the new language version.

The aim of the study is to translate and validate French versions of specific scales of QOL in peripheral facial palsy patients: FDI and FaCE. Secondary objective is to evaluate QOL of patients depending on PFP etiology.

Translation process will be done respecting internationally recognized rules. A pilot study will be performed on 5 physicians and 5 patients in order to validate the questionnaires translations. French versions obtained for these 2 questionnaires will be used for their validation on 80 patients suffering from PFP in our hospital.

Cronbach's alpha will be estimated to check internal consistency of FDI and FaCE scales. Test re-test reliability will be calculated with inter-class correlation, reiterating questionnaires one week later. Scores of FDI and FaCE scales will be compared to House-Brackmann and Sunnybrook clinical evaluation scales, estimating correlation coefficient. Social function of FDI and FaCE scales will also be compared with general scale SF-36 scores, estimating a correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Patient with peripheral facial palsy
* Age over 18 years old.
* Subject wishing and able to give informed consent and to respect the requirements of the protocol

Exclusion Criteria:

* Patient not being French.
* Patient who can not read French.
* Facial graduation.
* Facial dysfunction other than PFP such as facial trauma.
* Major medical or psychiatric illness that, in the opinion of the investigator, would pose a risk to the subject or could compromise compliance with the study protocol.
* Participation in other studies in the 30 days prior to inclusion in this study.
* Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
"Facial disability Index" (FDi) | one week
  questionnaire to assess the oral, ocular and the influence of facial impairment on emotions and daily activity

SECONDARY OUTCOMES:
Facial Clinimetric Evaluation" (FaCE) | one week
  questionnaire to asses facial deficit and disability relating to 6 areas: facial movement, facial comfort, oral function, ocular comfort, tear control and social function
House-Brackmann score | one week
  The House-Brackmann score is a score to grade the degree of nerve damage in a facial nerve palsy. The measurement is determined by measuring the upwards (superior) movement of the mid-portion of the top of the eyebrow, and the outwards (lateral) movement of the angle of the mouth. Each reference point scores 1 point for each 0.25 cm movement, up to a maximum of 1 cm. The scores are then added together, to give a number out of 8
Sunnybrook index | one week
  clinical evaluation calculating a score depending of Resting Symmetry, Symmetry of Voluntary Movement and Synkinesis
SF-36 score | one week
  The Short Form (36) Health Survey is a 36-item.
  It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — ASSISTANCE PUBLIQUE DES HOPITAUX DE MARSEILLE
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France